CLINICAL TRIAL: NCT04319861
Title: Long-term Clinical Results With the Use of an Anal Fistula Plug for the Treatment of Trans-sphincteric Anal Fistulas
Brief Title: Anal Fistula Plug, a Retrospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhen Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Plug 2020
Record Dates: First submitted 2020-03-15; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Healing Rate; Recurrence; Complication
Keywords: Anal fistula plug; Trans-sphincteric anal fistula; Overall healing rate; Anal function; Risk factors; Minimally invasive
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anal fistula plug (Experimental): The anal fistula plug procedure was performed as followings. A fistula probe was used to identify fistula tracts, and internal and external openings. Gentle mechanical debridement was performed with a blunt curette to remove the necrotic tissue with care not to enlarge the track, then hydrogen peroxide and sterile saline were used to repeatedly to irrigate the fistula. The anal fistutla plug was filled into the fistula, and sutured with a figure-of-eight 2-to-0 Vicryl suture to ensure the plug was fixed in the internal opening of the fistula, avoiding the anal fistula plug being extruded. Trimming the plug at the external fistula and the external opening was left open to ensure adequate drainage.
  Interventions: Procedure: Anal fistula plug procedure

INTERVENTIONS:
Procedure: Anal fistula plug procedure — A fistula probe was used to identify fistula tracts, and internal and external openings. Gentle mechanical debridement was performed with a blunt curette to remove the necrotic tissue with care not to enlarge the track, then hydrogen peroxide and sterile saline were used to repeatedly to irrigate the fistula. The anal fistutla plug was filled into the fistula, and sutured with a figure-of-eight 2-to-0 Vicryl suture to ensure the plug was fixed in the internal opening of the fistula, avoiding the anal fistula plug being extruded. Trimming the plug at the external fistula and the external opening was left open to ensure adequate drainage.

SUMMARY:
In this study, we retrospectively reviewed clinical data of patients who were treated with an anal fistula plug for trans-sphincteric anal fistulas, and evaluated the long-term therapeutic effect of an anal fistula plug and the risk factors impacting anal fistula healing. In addition, we assessed the effects of post-operative changes on anal function, as well as the risk factors affecting anal function.

DETAILED DESCRIPTION:
Treatment of anal fistulas, especially involving signiﬁcant anal sphincters, continues to represent a challenge for surgeons. Surgery has been the mainstay of treatment, and the ideal goal of anal fistula treatment is to obliterate the fistulous tract, while preserving the anal sphincter and avoiding fecal incontinence. The anal fistula plug is a sphincter-sparing procedure that uses biological substances to close an anorectal fistula. Several studies have preliminarily shown that the anal fistula plug had advantages of simple and repeatable application, preservation of sphincter integrity, minimal patient discomfort, and subsequent surgical options if needed. The healing rate of anal fistula plug varied widely, which range from 14% to 88%, and no significant effect on anal function in the short term. Therefore, long-term observation and a large sample size are needed to evaluate the long-term healing rate of an anal fistula plug, and the effect on anal function. The aim of this study is to assess the long-term therapeutic effect of an anal fistula plug in patients with trans-sphincteric fistula-in-ano, as well as the impact on anal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trans-sphincteric anal fistula.
* The case information was complete.
* Not receive other treatment previously.

Exclusion Criteria:

* Fistulas related to Crohn's disease, ulcerative colitis or anorectal tumors.
* Underwent surgical incision and drainage for acute perianal infections within 3 months.
* Multiple fistula tracts > 2.
* Poor underlying condition and unable to tolerate surgery.

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Healing rate | 8 years postoperatively
  The healing rate of anal fistula plug in 8 years postoperatively

SECONDARY OUTCOMES:
Anal function | 8 years postoperatively
  Cleveland Clinic Florida (Wexner) incontinence scale

CONTACTS AND LOCATIONS:
Overall Officials: Jiagang Han, Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No